CLINICAL TRIAL: NCT07072091
Title: Focusing the Shoulder or Considering the Whole-Body? A Randomized Controlled Trial on Physiotherapy Protocols for the Painful Shoulder in Volleyball Players
Brief Title: Focusing the Shoulder or Considering the Whole-Body in Volleyball Physiotherapy
Acronym: FocusVolley
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Trieste (Other)
Responsible Party: Principal Investigator, Alex Buoite Stella, PhD, Assistant professor, University of Trieste
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DSM_Fisio_SpallaPallavolo25
Record Dates: First submitted 2025-05-30; First posted 2025-07-18 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Shoulder Pain; Volleyball Players
MeSH Terms: conditions — Shoulder Pain | interventions — Educational Status

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy controls (No Intervention): A convenience sample of healthy volleyball players for cross-sectional comparison
- Total body physiotherapy group (Experimental): Physiotherapy intervention consisting in whole body exercise and treatment
  Interventions: Other: Total body physiotherapy
- Focus shoulder group (Active Comparator): Physiotherapy intervention consisting in shoulder exercise and treatment
  Interventions: Other: Focus shoulder physiotherapy
- No physiotherapy group (Other): No physiotherapy, only education
  Interventions: Other: Education

INTERVENTIONS:
Other: Total body physiotherapy — This intervention consists in 5 weeks of 2 x week 60 min sessions of physiotherapy consisting in active exercise performed in upper limb, trunk, and lower limb muscles, in a whole-body approach.
  Arms: Total body physiotherapy group
Other: Focus shoulder physiotherapy — This intervention consists in 5 weeks of 2 x week 60 min sessions of physiotherapy consisting in active exercise performed only in the shoulder district, focusing on the trunk-arm muscles.
  Arms: Focus shoulder group
Other: Education — Single education session providing information about posture hygiene and proper warm-up
  Arms: No physiotherapy group

SUMMARY:
Shoulder pain can be common in overhead sports, and in particular, in volleyball. Different physiotherapy protocols can be adopted depending on the suspected pathophysiological mechanisms. Despite most of the protocols rely only on the shoulder district, some research suggests that treating the whole-body might produce better results as it could influence kinematic chains and correct muscle imbalances. The aim of this study will be to compare the effects of two physiotherapy protocols (shoulder focus or whole body) compared to only education without physiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* practicing volleyball for at least 5 years with a training volume of minimum 5 h/wk

Exclusion Criteria:

* history of previous surgical intervention or fractures on the shoulder or spine

Ages: 17 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07-20 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Isometric strength with handheld dynamometer (Newtons) | At enrollment and at the end of treatment at 5 weeks
  Isometric strength during shoulder flexion, extension, external and internal rotation, bilaterally

SECONDARY OUTCOMES:
Lateral symmetry (%) | At enrollement and at the end of treatment after 5 weeks
  Lateral symmetry will be assessed as percentage between the two upper limbs for the investigated muscles (pectoralis major, latissimus dorsi, upper trapezius, middle trepezius, lower trapezius, anterior deltoid, posterior deltoid) using the tensiomyography system
Time of contraction (ms) | At enrollement and at the end of treatment after 5 weeks
  Time of contraction (ms), i.e. the time requiring the muscle to reach the peak of muscle displacement, will be assessed as percentage between the two upper limbs for the investigated muscles (pectoralis major, latissimus dorsi, upper trapezius, middle trepezius, lower trapezius, anterior deltoid, posterior deltoid) using the tensiomyography system
Muscle belly displacement (mm) | At enrollement and at the end of treatment after 5 weeks
  Muscle belly displacement (mm), i.e. the amplitude of muscle displacement, will be assessed as percentage between the two upper limbs for the investigated muscles (pectoralis major, latissimus dorsi, upper trapezius, middle trepezius, lower trapezius, anterior deltoid, posterior deltoid) using the tensiomyography system

CONTACTS AND LOCATIONS:
Locations (1):
- University of Trieste - Exercise Physiology and Kinesiology Lab, Trieste, Trieste, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jones SD Jr, Safran MR. Current concepts: the hip, core and kinetic chain in the overhead athlete. J Shoulder Elbow Surg. 2024 Feb;33(2):450-456. doi: 10.1016/j.jse.2023.10.009. Epub 2023 Nov 23. PMID 38007174
- [Background] Erkan R, Telci EA. Impact of Stabilization Exercises on Athletic Performance and Injury Risk in College Volleyball Players. Int J Sports Physiol Perform. 2025 May 13;20(7):948-957. doi: 10.1123/ijspp.2024-0348. Print 2025 Jul 1. PMID 40360147